CLINICAL TRIAL: NCT07024212
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of DR10624 Injection in Subjects at High Risk of Liver Fibrosis With Metabolic Dysfunction-associated Steatotic Liver Disease and Metabolic Dysfunction and Alcohol Associated Steatotic Liver Disease
Brief Title: Phase II Study Evaluating the Efficacy and Safety of DR10624 Injection in MASLD and MetALD Subjects
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Doer Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DR10624-202
Record Dates: First submitted 2025-04-24; First posted 2025-06-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: MASLD
Keywords: NASH; MASH; NAFLD; MAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1：DR10624 injection/Placebo (SC, qw) (Experimental): DR10624 injection/Placebo (SC, qw)
  Interventions: Drug: DR10624 Injection; Drug: Placebo
- Cohort 2：DR10624 injection/Placebo (SC, qw) (Experimental): DR10624 injection/Placebo (SC, qw)
  Interventions: Drug: DR10624 Injection; Drug: Placebo
- Cohort 3：DR10624 injection/Placebo (SC, qw) (Experimental): DR10624 injection/Placebo (SC, qw)
  Interventions: Drug: DR10624 Injection; Drug: Placebo
- Cohort 4：DR10624 injection/Placebo (SC, qw) (Experimental): DR10624 injection/Placebo (SC, qw)
  Interventions: Drug: DR10624 Injection; Drug: Placebo
- Cohort 5：DR10624 injection/Placebo (SC, qw) (Experimental): DR10624 injection/Placebo (SC, qw)
  Interventions: Drug: DR10624 Injection; Drug: Placebo

INTERVENTIONS:
Drug: DR10624 Injection — Drug: DR10624 injection
Drug: Placebo — Drug: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, Phase II clinical trial that consists of two parts. The primary objective of Part 1 is to assess the preliminary efficacy of DR10624 Injection in MASLD subjects at high risk of liver fibrosis. The secondary objectives are to assess the safety and tolerability, PK profiles, and immunogenicity of DR10624 Injection in these subjects. The exploratory objectives are to assess the efficacy of DR10624 Injection in these subjects using LSM assessed by MRE, and its impact on Lp(a) and body composition.The primary objective of Part 2 is to assess the safety and tolerability of DR10624 Injection in MetALD subjects at high risk of liver fibrosis. This clinical trial is currently only conducting Part 1 of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have signed the informed consent form before the trial, and fully understood the trial content, process and possible adverse reactions;
2. Males or females aged 18-75 years (inclusive) at the time of signing the informed consent form;
3. LFC ≥ 10% assessed by MRI-PDFF (MRI-PDFF results that are obtained at the study site within 6 weeks prior to randomization are acceptable);
4. Screening FibroScan® with liver stiffness (LSM): ≥ 8 Kpa, and < 15 Kpa;
5. Have a body mass index (BMI) between 25.0 and 40.0 kg/m2 (inclusive) at screening;
6. Less than 5% change in body weight within 6 months prior to randomization;
7. If there is a history of type 2 diabetes, a stable treatment regimen must be maintained for at least 12 weeks prior to screening;
8. Females of childbearing potential and males must agree to use effective contraception during the study and for a specified period after the last dose of the investigational medicinal product (2 months for females, 3 months for males).

Exclusion Criteria:

1. Presence of cirrhosis on liver biopsy or imaging results, or have a history of cirrhosis;
2. Other causes of liver disease based on medical history and/or laboratory tests;
3. Previous (within 5 years before randomization) or planned (during the study period) obesity treatment with metabolic surgery or device-based therapy subjects with reversible weight-loss devices removed more than 12 months prior to randomization are eligible;
4. Type 1 diabetes;
5. History of malignancies within the last 5 years prior to screening, or malignancies that occurred more than 5 years ago but which are still currently active. Local squamous cell carcinoma of the skin or cervical intraepithelial neoplasia that has been cured without signs of recurrence is acceptable;
6. Presence of severe or uncontrolled underlying disease that, in the opinion of the investigator, renders the subject unsuitable for treatment with the investigational medicinal product or unable to complete study, or is likely to interfere with the evaluation of study results;
7. Subjects who have a history of bone trauma, fracture, or bone surgery within 2 months prior to screening, or concomitant bone disorders such as osteomalacia or known, untreated severe vitamin D deficiency (serum 25-hydroxyvitamin D ≤5 ng/mL); or a T-score ≤-2.5 for bone mineral density measured by DXA in the axial skeleton (lumbar vertebrae 1-4, femur neck, or total hip);
8. Subjects who have a history of medullary thyroid carcinoma, multiple endocrine neoplasia type 2, or a related family history;
9. Any significant abnormal laboratory findings from screening to randomization;
10. Subjects who have used or plan to use the following medications that may cause steatosis/steatohepatitis cumulatively for ≥4 weeks within 24 weeks prior to randomization or during the study: amiodarone, methotrexate, systemic corticosteroids (dose >5 mg/day prednisone equivalent), estrogens (dose greater than that used for hormone replacement therapy or contraception), tetracyclines, tamoxifen, anabolic steroids, valproic acid, or other drugs known to have hepatotoxicity, etc.;
11. Use of any of the following medications cumulatively for ≥4 weeks within 24 weeks prior to randomization or planned during the study: high-dose vitamin E (daily dose >400 IU), obeticholic acid, pioglitazone, berberine, or thyroid hormones (subjects with hypothyroidism who have received stable replacement therapy for at least 3 months prior to randomization are acceptable), etc.;
12. Use of antidiabetic drugs other than metformin, sulfonylureas, alpha-glucosidase inhibitors, glucokinase activators (GKA), or sodium-glucose cotransporter 2 (SGLT-2) inhibitors within 12 weeks prior to screening or planned during the study;
13. Use of Schisandra preparations (e.g., bifendate, bicyclol) within 6 weeks prior to randomization, or use of the following hepatoprotective drugs (including but not limited to reduced glutathione, glucuronolactone, glycyrrhizic acid preparations, polyene phosphatidylcholine, ursodeoxycholic acid, nicotinamide, liver-protecting tablets, silymarin, etc.) or other hepatoprotective Chinese proprietary medicines or health products within 2 weeks prior to randomization; or planned use of such drugs during the study;
14. Use of weight-loss drugs such as orlistat or GLP-1 receptor agonists, or other drugs with the same target as the investigational medicinal product [e.g., fibroblast growth factor-21 (FGF21) analogs, glucagon receptor (GCGR) agonists, etc.], within 6 weeks prior to screening or planned during the study;
15. Use of anti-tumor necrosis factor α (TNF-α) drugs, such as adalimumab or etanercept, etc., within 6 weeks prior to screening or planned during the study;
16. Known or suspected intolerance or hypersensitivity to the investigational medicinal product or any of its excipients; or known intolerance or hypersensitivity to drugs with the same target (e.g., FGF21 analogs, GLP-1 receptor agonists, GCGR agonists, etc.);
17. Subjects who have participated in clinical trials of other drugs and used investigational medicinal product within 12 weeks or 5 half-lives (whichever is longer) prior to screening, or those who have participated in medical device or vaccine clinical trials;
18. Alcohol consumption for at least 12 consecutive weeks within 1 year prior to screening, defined as any of the following: > 210 grams of ethanol per week for males on average, > 140 grams per week for females on average;
19. History of drug abuse or use of illicit drugs within 3 years prior to screening;
20. Pregnant or breastfeeding females, or females with a positive serum pregnancy test prior to randomization;
21. Subjects who, in the investigator's opinion, are otherwise not suitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Changes of LFC | From baseline to Week 12
  Relative percentage changes (%) of Liver Fat Content (LFC) from baseline to Week 12, assessed by MRI-PDFF.

SECONDARY OUTCOMES:
Changes of Controlled Attenuation Parameter (CAP) | From baseline to Week 12
  Changes of CAP from baseline to Week 12, assessed by FibroScan® VCTE.
Changes of Liver Stiffness Measurement (LSM) | From baseline to Week 12
  Changes of LSM from baseline assessed by FibroScan® VCTE.
Changes of LFC | From baseline to Week 12
  Changes of LFC from baseline to Week 12, assessed by MRI-PDFF.
Proportion of subjects achieving a relative reduction of LFC | From baseline to Week 12
  Proportion of subjects who achieve a relative reduction of LFC by ≥30%, ≥50%, or ≥70% from baseline to Week 12.
Proportion of subjects with LFC <5% | From baseline to Week 12
  Proportion of subjects with LFC <5% after 12 weeks of treatment.
Changes of liver enzymes | From baseline to Week 16
  Changes of liver enzymes from baseline to Week 16.
Proportion of subjects with ≥17 U/L reduction of ALT | From baseline to week 16
  Proportion of subjects with ≥17 U/L reduction of ALT from baseline to Week 16.
Changes of glucose metabolism-related parameters | From baseline to Week 12
  Changes of glucose metabolism-related parameters from baseline to Week 12.
Changes of lipid profiles | From baseline to Week 16
  Changes of lipid profiles from baseline to Week 16.
Changes of body weight | From baseline to Week 16
  Changes of body weight from baseline to Week 16
Changes of BMI | From baseline to Week 16
  Changes of BMI from baseline to Week 16, BMI = weight (kg)/height2 (m2), height is measured only at screening, while weight is measured at each corresponding visit.
Changes of hip circumference | From baseline to Week 16
  Changes of hip circumference from baseline to Week 16. The hip circumference should be recorded in cm, accurate to mm (e.g., 96.6 cm).
Changes of waist-to-hip ratio | From baseline to Week 16
  Changes of waist-to-hip ratio from baseline to Week 16 Waist-to-hip ratio = waist circumference (cm) / hip circumference (cm).
Changes of fibrosis biomarkers | From Baseline to Week 12
  Changes from baseline in fibrosis biomarkers.
Changes of hepatic inflammation markers | From baseline to week 12
  Changes of hepatic inflammation markers from baseline to Week 12
Analysis of Safety Endpoints | From baseline to week 16
  Safety parameters from baseline to Week 16
Immunogenicity analysis | From baseline to Week 16
  Assess the immunogenicity from baseline to Week 16
Pharmacokinetics profiles of DR10624 Injection | From baseline to Week 12
  Measurement of DR10624 plasma concentration and calculation of C trough.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Wai-Sun Wong, M.D., Study Chair — Prince of Wales Hospital, The Chinese University of Hong Kong; Junping Shi, M.D., Principal Investigator — The Affiliated Hospital of Hangzhou Normal University
Locations (4):
- China (3):
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - The First Hospital of Jilin University, Changchun
  - Nanjing Gulou Hospital, Nanjing
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong, Hong Kong